CLINICAL TRIAL: NCT04011358
Title: Retinal Vein Occlusion and Obstructive Sleep Apnea: A Case Control Study
Acronym: SASOVR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Given the health context and the work overload, this study will not be possible. We therefore abandon this project
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHRO-2018-14
Record Dates: First submitted 2019-06-07; First posted 2019-07-08 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Retinal Vein Occlusion; Obstructive Sleep Apnea
Keywords: Retinal Vein Occlusion; central retinal vein occlusion; branch retinal vein occlusion; obstructive sleep apnea; sleep apnea
MeSH Terms: conditions — Retinal Vein Occlusion; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: case-control comparison study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Other): Patient with Retinal Vein Occlusion
  Interventions: Other: Sleeping Monitor
- Patient control (Other): Patient with no Retinal Vein Occlusion
  Interventions: Other: Sleeping Monitor

INTERVENTIONS:
Other: Sleeping Monitor — to evaluate obstructive sleep apnea

SUMMARY:
This study purpose is to evaluate the association between Retinal Vein Occlusion and Obstructive Sleep Apnea.

DETAILED DESCRIPTION:
There will be two groups of 50 patients. One with Retinal Vein Occlusion, and the other one, with no Retinal Vein Occlusion will be chosen from the consultation.

The compared group will be paired on different criteria including hypertension, ocular hypertension, diabetes, sex, age.

They will all spend a night at home with a Sleeping Monitor (Nox T3) in order to evaluate if they have an Obstructive Sleep Apnea.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an Retinal Vein Occlusion for one group (patients)
* All patients with no Retinal Vein Occlusion for the other group (control)

Non-inclusion Criteria:

* minor
* Severe Insomnia
* Neuromuscular Disease with respiratory muscle impairment
* Chronic opioid medication
* Pregnancy women.
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea index >5/hour | Hour 12
  Obstructive Sleepin Apnea diagnostic depends only on the AHI which is measured by the Sleeping Monitor at home.

SECONDARY OUTCOMES:
Berlin Questionnaire sleep test | Hour 12
  High Risk of Sleep Apnea Syndrome:
  If there are 2 or more Categories where the score is 2 or above
  Low Risk of Sleep Apnea Syndrome:
  If there is only 1 or no Categories where the score is 2 or above

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BONICEL, Dr, Principal Investigator — CHR Orléans
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Glacet-Bernard A, Leroux les Jardins G, Lasry S, Coscas G, Soubrane G, Souied E, Housset B. Obstructive sleep apnea among patients with retinal vein occlusion. Arch Ophthalmol. 2010 Dec;128(12):1533-8. doi: 10.1001/archophthalmol.2010.272. PMID 21149775
- [Result] Chou KT, Huang CC, Tsai DC, Chen YM, Perng DW, Shiao GM, Lee YC, Leu HB. Sleep apnea and risk of retinal vein occlusion: a nationwide population-based study of Taiwanese. Am J Ophthalmol. 2012 Jul;154(1):200-205.e1. doi: 10.1016/j.ajo.2012.01.011. Epub 2012 Mar 30. PMID 22464364
- [Result] Kwon HJ, Kang EC, Lee J, Han J, Song WK. Obstructive Sleep Apnea in Patients with Branch Retinal Vein Occlusion: A Preliminary Study. Korean J Ophthalmol. 2016 Apr;30(2):121-6. doi: 10.3341/kjo.2016.30.2.121. Epub 2016 Mar 25. PMID 27051260
- [Result] Agard E, El Chehab H, Vie AL, Voirin N, Coste O, Dot C. Retinal vein occlusion and obstructive sleep apnea: a series of 114 patients. Acta Ophthalmol. 2018 Dec;96(8):e919-e925. doi: 10.1111/aos.13798. Epub 2018 Sep 6. PMID 30188014